CLINICAL TRIAL: NCT04037605
Title: Hormonal Mechanisms of Sleep Restriction - Axis Study in Older Men and Postmenopausal Women
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Peter y. Liu, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: P31056-01R
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sleep Restriction
Keywords: Testosterone; Cortisol
MeSH Terms: interventions — Ketoconazole; ganirelix; Dexamethasone; Calcium Dobesilate; Luteinizing Hormone, beta Subunit; Hydrocortisone; hydrocortisone hemisuccinate; Gonadotropin-Releasing Hormone; Corticotropin-Releasing Hormone; corticorelin ovine; Saline Solution; Injections

STUDY DESIGN:
Intervention Model Description: Blood is sampled every 10 minutes from 4 pm to 9 pm for future mathematical deconvolution in order to determine hormone pulse characteristics in response to the clamp conditions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 3 of the 4 conditions are masked by use of identical injections and pills. However one condition (adrenal testis) is not masked. Hence the study is partially masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control Condition (Experimental): 8 am - Saline Solution for Injection
  10 am - Placebo oral capsule
  1 pm - Saline Solution for Injection
  4 pm - Placebo oral capsule & start hourly blood sampling
  7 pm- Gonadorelin (GnRH) and Corticorelin (CRH) injections
  9 pm - Saline Solution for Injection & last blood sample
  Interventions: Drug: Gonadorelin (also known as Lutrepulse); Drug: Corticorelin (also known as Acthrel); Drug: Placebo oral tablet; Drug: Saline Solution; Drug: Saline solution for injection
- Hypothalamic Condition (Experimental): 8 am -Ganirelix
  10 am - Placebo oral capsule
  1 pm - Dexamethasone injection
  4 pm- Placebo oral capsule and start of hourly blood sampling
  7 pm - GnRH and CRH injections
  9 pm - Saline Solution for Injection and last sample blood sample
  Interventions: Drug: Ganirelix; Drug: Dexamethasone injection; Drug: Gonadorelin (also known as Lutrepulse); Drug: Corticorelin (also known as Acthrel); Drug: Placebo oral tablet; Drug: Saline solution for injection
- Pituitary Condition (Experimental): 8 am - Saline Solution for Injection
  10 am - Ketoconazole Pill
  1 pm - Saline Solution for Injection
  4 pm - Ketoconazole Pill & start of hourly blood sampling
  7 pm - GnRH and CRH
  9 pm - Hydrocortisone Injection and last blood sample
  Interventions: Drug: Ketoconazole Pill (also known as nizoral); Drug: Hydrocortisone Injection (also known as solu-cortef); Drug: Gonadorelin (also known as Lutrepulse); Drug: Corticorelin (also known as Acthrel); Drug: Saline Solution
- Adrenal/Testis Condition (Experimental): 10 pm - Ganirelix Injection & Dexamethasone Pills (night before)
  8 am - Start of hourly blood sampling
  10 am - Dexamethasone Pills
  11 am - Last hourly blood sample taken
  11:30 am - Start of blood sampling every 10 minutes
  1 pm - Recombinant Human Luteinizing Hormone (rhLH) Injection
  3 pm - rhLH Injection
  5 pm - rhLH Injection
  5 pm - Cosyntropin Injectable product
  7 pm - GnRH and CRH Injections
  9 pm - Last blood sample
  Interventions: Drug: Ganirelix; Drug: Dexamethasone Pill; Drug: Cosyntropin Injectable Product; Drug: Recombinant Human Luteinizing Hormone (also known as luveris); Drug: Gonadorelin (also known as Lutrepulse); Drug: Corticorelin (also known as Acthrel)

INTERVENTIONS:
Drug: Ketoconazole Pill (also known as nizoral) — Ketoconazole pill is taken 4 times per inpatient visit
  Arms: Pituitary Condition
Drug: Ganirelix — Ganirelix subcutaneous injection is administered twice per inpatient visit
  Arms: Adrenal/Testis Condition; Hypothalamic Condition
Drug: Dexamethasone Pill — Dexamethasone pills is taken twice per inpatient visit
  Arms: Adrenal/Testis Condition
Drug: Dexamethasone injection — Dexamethasone IV injection is given twice per inpatient visit
  Arms: Hypothalamic Condition
Drug: Cosyntropin Injectable Product — Cosyntropin injection is given twice per inpatient visit
  Arms: Adrenal/Testis Condition
Drug: Recombinant Human Luteinizing Hormone (also known as luveris) — Recombinant Human Luteinizing Hormone is given as 6 IV infusion pulses per inpatient visit
  Arms: Adrenal/Testis Condition
Drug: Hydrocortisone Injection (also known as solu-cortef) — Hydrocortisone IV push is given twice per inpatient visit
  Arms: Pituitary Condition
Drug: Gonadorelin (also known as Lutrepulse) — Gonadorelin IV injection is given twice per inpatient visit
Drug: Corticorelin (also known as Acthrel) — Corticorelin IV injection is given twice per inpatient visit
Drug: Placebo oral tablet — Placebo for Ketoconazole are given 4 times per inpatient visit
  Arms: Control Condition; Hypothalamic Condition
Drug: Saline Solution — Saline Solution (Placebo) for Dexamethasone IV injection or hydrocortisone IV injection given up to four times per inpatient visit
  Arms: Control Condition; Pituitary Condition
Drug: Saline solution for injection — Saline Solution (placebo) for ganirelix subcutaneous injection
  Arms: Control Condition; Hypothalamic Condition

SUMMARY:
The purpose of this study is to 1) determine how hypothalamic-pituitary-adrenal axis (HPA axis) activation occurs with sleep restriction and 2) evaluate how hypothalamic-pituitary-gonadal axis (HPG axis) deactivation occurs with sleep restriction. The investigator will also examine the cognitive function associated with sleep restriction, including food intake and food cravings.

DETAILED DESCRIPTION:
Sleep restriction and its consequences are major public health problems, especially in older adults. Among the more severe physiological sequelae of sleep restriction is the development of insulin resistance. The mechanisms by which sleep restriction leads to increased insulin resistance are unknown, especially in vulnerable older adults; such research informs development of targeted interventions against the sleep loss/insulin resistance link.

This study will administer drugs to clamp the function of each of these nodes to determine the regulatory changes that have occurred with sleep restriction. Even though the study is randomized order in design, the main comparison is before and after sleep restriction under each of these clamp conditions. Participants are admitted to the chronobiology laboratory where they are given 1 night of 10 hours sleep opportunity, followed by 4 nights of 4 hours sleep opportunity.

Up to 40 participants can be enrolled. However, participants will be allowed an opportunity to be randomized to all 4 conditions so that as few as 10 participants may be required. We anticipate 5 men and 5 women will be enrolled assuming each undergoes all 4 clamp conditions.

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal women aged 60-80 years
* Willingness to provide written informed consent
* Stable weight over preceding 6 weeks
* Body Mass index (BMI) 22-28 kg/m2
* Physically and psychologically healthy
* Good habitual sleep with regular bedtimes
* Neither extreme morning- nor extreme evening-type using Horne-Ostberg Morningness-Eveningness criteria

Exclusion Criteria:

* Medications that interfere with the adrenal or gonadal axis will be excluded
* Unable or unwilling to provide IRB (Internal Review Board)-approved informed consent
* Clinical disorders and/or illnesses
* Current medical or drug treatment, as assessed by questionnaire
* History of brain injury or of learning disability
* Vision or hearing impairment unless corrected back to normal
* Anemia (Hct <38%)
* History of psychiatric illness
* Clinically significant abnormalities in blood and urine, and free of traces of drugs
* Other endocrine abnormalities including hypothyroidism or adrenal failure; primary gonadal disease as indicated by serum LH (luteinizing hormone) or FSH (follicle stimulating hormone) concentration >10 or >15 IU/L, respectively, hyperprolactinemia indicated by prolactin >25ug/L
* Type 2 Diabetes (HgbA1C)
* Current smoker
* Recent or concurrent drug or alcohol abuse
* Blood donation in previous eight weeks
* Travel across time zones within one month of entering the study
* Sleep or circadian disorder
* Shift work within three months of entering the study
* Irregular bedtimes (not between 6 and 10 hours in duration)
* Unoperated obstructive uropathy, recurrent prostatitis, indeterminate prostatic nodularity, Hx or Suspicion of cancer of the prostate gland or PSA (prostate-specific antigen) >4ng/ml
* Previous adverse reaction to sleep deprivation or any of the drugs to be administered
* Concurrent participation in another research study
* Mini- mental state examination (MMSE) < 27

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Average Blood Cortisol Concentration | 5 days
  Cortisol is measured in blood every 10 minutes for a 5 hour period, at the beginning and at the end of 4 nights of sleep restriction. The average cortisol is the parameter of interest.
Average Blood Testosterone Concentration | 5 days
  Testosterone is measured in blood every 10 minutes for a 5 hour period, at the beginning and at the end of 4 nights of sleep restriction. The average cortisol is the parameter of interest.

SECONDARY OUTCOMES:
Peak Blood Cortisol Concentration | 5 days
  This is the single maximal blood cortisol concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Peak Blood Testosterone Concentration | 5 days
  This is the single maximal blood testosterone concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Trough Blood Cortisol Concentration | 5 days
  This is the single minimal blood cortisol concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Trough Blood Testosterone Concentration | 5 days
  This is the single minimal blood testosterone concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Reaction time on Psychomotor Vigilance Task | 5 days
  This is measured by lapses in attention. As the person becomes more sleepy, there are more lapses (reaction time >500 ms), at the beginning and at the end of 4 nights of sleep restriction.
Karolinska Sleepiness Scale | 5 days
  Measures how sleepy participants are using a scale of 1 (extremely alert) through 9. This scale will be used to assess changes in sleepiness throughout the day and through 4 nights of sleep restriction.
Two card gambling task | 5 days
  Computerized neurobehavioral testing to determine how 4 nights of sleep restriction affects participants' decision making. The end point is discriminability index, d'.
Modified Sternberg working memory test | 5 days
  Computerized neurobehavioral testing to determine how 4 nights of sleep restriction affects reaction time and accuracy.
Caloric Intake | 5 days
  The food given to participants is weighed. The amount that is not consumed is also weighed. The difference in weight is the amount of calories consumed.
Hunger | 5 days
  Hunger levels are assessed using the Flint visual analogue scale (VAS) to assess how 4 nights of sleep restriction affects participants' appetite.The Flint VAS asks the participant to rate 8 aspects of their hunger level on a scale from 1-5.
Food Cravings | 5 days
  Food cravings are measured using the Food Cravings Index (FCI) scale to assess which food groups each participant has cravings for and how their cravings change during 4 nights of sleep restriction. The participant ranks their craving for 33 food items on a scale from 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MD, PhD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No